CLINICAL TRIAL: NCT06952582
Title: Effect of Information-motivation-behavioral Skill Model-based Safer Sexual Dual Protection Intervention on Knowledge, Motivation, Behavioral Skills and Practice of Abstinence and Dual Protection Use Among Female University Students in Ethiopia: A Quasi-experimental Study
Brief Title: Promoting Safer Sexual Dual Protection Behaviors for Female University Students to Reduce Risks of Both STI/HIV and Unintended Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jimma University (Other)
Responsible Party: Principal Investigator, Banti Negero Feyisa, Masters of Public Health in Reproductive Health, Jimma University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Bonsakoo2003&Ebanufbanti2009
Record Dates: First submitted 2025-04-20; First posted 2025-05-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Sexually Transmitted Infections(STIs); HIV/AIDS; Unintended Pregnancy
Keywords: IMB model,; HIV risk reduction,; Safer sexual dual protection behaviors,; Dual protection use
MeSH Terms: conditions — Sexually Transmitted Diseases; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: On the basis of elicitation research findings, the IMB model-based safer sexual dual protection intervention was designed to promote safer sexual dual protection behaviors, including abstinence and dual protection use, for both sexually inexperienced and sexually experienced female university students to reduce the risk of both STI/HIV and unwanted pregnancy. Participants in intervention group will receive the IMB model-based safer sexual dual protection education, while participants in control group will receive the usual standard HIV education.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): The control group will only receive the usual standard HIV education programs for university students.
- Safer sexual dual protection (SSDP) intervention (Experimental): The intervention group will receive the IMB model-based safer sexual dual protection intervention designed to promote safer sexual dual protection behaviors, including abstinence and dual protection use, for both sexually inexperienced and sexually experienced female university students to reduce the risk of both STI/HIV and unwanted pregnancy.
  Interventions: Behavioral: The IMB model-based safer sexual dual protection educational intervention

INTERVENTIONS:
Behavioral: The IMB model-based safer sexual dual protection educational intervention — The IMB model based safe sexual dual protection education was designed to provide factual information about sexual risks of STI/HIV and unwanted pregnancy and the benefits of safer sexual dual protection behaviors including abstinence and dual protection use, enhance motivation to practice primary sexual abstinence for sexually inexperienced youth and dual protection use for sexually experienced young women, and teach specific behavioral skills required for practicing abstinence and/or negotiate safer sex with partners to use condoms/dual protection for simultaneous prevention of both risks of STI/HIV and unwanted pregnancy among youth at risk.
  Arms: Safer sexual dual protection (SSDP) intervention

SUMMARY:
Background: Young women are at the greatest risk for STI/HIV infections and unintended pregnancy resulting from unsafe sexual practices. While there is a growing interest in promoting dual protection as a means of preventing both risks of HIV/STIs and unwanted pregnancy simultaneously, there is limited evidence of effective interventions and strategies for promoting dual protection behaviors in youth based on theoretical models. This study aimed to evaluate the effectiveness of an information-motivation-behavioral skills (IMB) model-based safer sexual dual protection (SSDP) intervention to promote safer sexual dual protection behaviors among female university students in Ethiopia.

Methods: We conducted a quasi-experimental nonrandomized control group design with a pretest-posttest study to assess changes in the levels of knowledge, motivation, behavioral skills, and practice of safe sexual dual protection behaviors with dual protection use in the intervention group compared to the control group. We recruited 1,020 female university students from two campuses of Mattu University using non-randomized assignment of each campus to either the intervention group or the control group. We collected data from both groups using a self-administered questionnaire at baseline and six months post-intervention. At both times, the collected data were cleaned, edited, and analyzed using SPSS version 23. For the baseline data analysis, we used descriptive statistics to summarize the distribution of participants based on their demographic characteristics and levels of information, motivation, behavioral skills, and behaviors. We also conducted bivariate and multivariate analyses using Structural Equation Modeling (SEM) with AMOS 23 (Teo, 2009; Kline, 2023) to examine correlates and predictors of risky and safer sexual practices and dual protection use and identify important variables to be addressed in targeted intervention for this population. Then, based on the elicitation research findings, we designed IMB-model-based SSDP interventions consisting of 16-hrs sessions to be delivered over a 6 weeks period. To evaluate the intervention effects at posttest, we performed a series of statistical analyses, such as chi-square (χ2) tests of differences between the two groups, along with 95% CI for the differences, and logistic regression analysis of the intervention effects, along with AOR for the effect size measure, after controlling for the effects of other confounding variables.

DETAILED DESCRIPTION:
Introduction The dual burden of HIV/AIDS and unwanted pregnancy continues to be a major public health concern worldwide, with young women disproportionately affected. In 2020, of the estimated 1.5 of people newly infected with HIV worldwide, approximately 260,000 were adolescent girls and young women aged 15--24 years, 83% of whom were in sub-Saharan Africa. In Ethiopia, although the adult HIV prevalence rate declined from 1.5% in 2011 to 0.93% in 2019, women remained disproportionately affected compared with men (1.22% vs. 0.64%), and the highest prevalence was observed among unmarried young women (9%). In addition, the rates of unwanted pregnancies among young women in Ethiopia remain high, with approximately 37% of unwanted pregnancies occurring among young women aged 20--24 years.

In response to the HIV epidemic, many HIV/AIDS prevention programs have emphasized safer sexual practices, such as abstinence, mutual monogamy, and condom use, as effective strategies for reducing the risk of HIV infection among youth. In addition, because young women are at increased risk and vulnerable to STI/HIV and unwanted pregnancy from unsafe premarital sex, and both can be prevented simultaneously be the same safer sexual practices as dual protection, the recent WHO/UNAIDS recommendation on HIV prevention for young women emphasizes the need for dual protection: defined as safer sexual behaviors that provide simultaneous protection against both HIV/STI and unwanted pregnancy through abstinence, consistent condom use, or dual-method use as complementary strategies for youth in settings with high HIV burden.

To achieve the maximum preventive effects, condoms are the only barrier method available to reduce the risk of STI/HIV infections and prevent pregnancy when used correctly and consistently, either alone or with other contraceptive methods as a dual protection among sexually active young women. Abstinence is the only sure way and most effective (100%) to avoid the risks of both HIV/STIs and unwanted pregnancy among unmarried youth who choose to remain abstinent. However, although trends in the use of contraceptive methods among unmarried sexually active young women in Ethiopia increased to 55% in 2016, only 4% used condoms, indicating that they were not dually protected and thus remained at an increased risk of HIV infection. Despite dual protection options for youth, there is limited evidence of effective interventions and strategies for promoting dual protection for youth in Ethiopia.

To date, school-based comprehensive sexuality education (CSE) has been considered the most effective strategy for protecting youth from the risk of HIV/STI and unwanted pregnancy by improving knowledge, attitudes, skills, and behaviors, such as delay of sexual debut, condom use, and contraceptive use. However, while young women may also need dual protection options to simultaneously prevent both risks of HIV/STIs and unwanted pregnancy, most of the existing sexual health education curriculum makes no explicit reference to dual protection messages for youth and thus remains unknown and not practiced. In addition, it is clear from research that for sexual health education intervention to be more effective in promoting sexual health behavior change, it must be guided by appropriate theoretical models for the development, implementation, and evaluation of the programs. Evidence from intervention studies indicates that theoretically derived and empirically based interventions can successfully promote the adoption of protective sexual behaviors among youth.

Theoretical perspectives Various behavioral theories have been applied to understand HIV risk behaviors and to promote safer sexual behaviors. Information-motivation-behavioral skills model is one that has been widely used in the areas of HIV prevention and received considerable attention and support for its comprehensiveness, specification of relationships, and ease of translating into targeted interventions to promote HIV prevention behaviors. The IMB model asserts that information, motivation, and behavioral skills are fundamental determinants of HIV-preventive behaviors. The model specifies that information and motivation work through behavioral skills to indirectly affect HIV-preventive behaviors. The model also assumes that information and motivation may have a direct effect on preventive behavior when complicated behavioral skills are not necessary for practice, such as abstinence, as opposed to using condoms by sexually active young women.

The IMB model's constructs are also regarded as a highly generalizable approach to understanding and promoting sexual health behaviors across populations and behaviors of interest. Within the IMB model, it is assumed that specific information, motivation, and behavioral skills can be most relevant to specific preventive practices, such as abstinence and condom use, within specific populations. Thus, the IMB model suggests that specification of the information, motivation, and behavioral skills content most relevant to the practice of a specific preventive behavior (abstinence and condom use) and identification of the IMB model's constructs that most powerfully influence the practice of preventive behavior are crucial to the design of effective conceptually and empirically targeted prevention interventions for specific populations. However, despite the recommendation for its application to a range of sexual health behaviors across populations and behaviors of interest, there is limited research using the IMB model to understand and promote safer sexual dual protection behaviors with dual protection use among young women at risk of STI/HIV infection and unwanted pregnancy. To fill these gaps, this study aimed to evaluate the effectiveness of an IMB model-based safer sexual dual protection intervention to improve levels of knowledge, motivation, behavioral skills, and practice of safer sexual dual protection behaviors, including abstinence and dual protection use, among female university students in Ethiopia.

Significance of the study:

Given that there is an increased risk and vulnerability of young women to STI/HIV and unwanted pregnancy from unsafe sex practice, and both can be prevented simultaneously by the same safer sexual practices as dual protection, understanding patterns and predictors of risky sexual practices and promoting safer sexual dual protection behaviors using theoretical models is essential for improving sexual and reproductive health of youth in settings with high HIV burden. Thus, by focusing on the application of the IMB model to promote safer sexual dual protection behaviors among youth, this study provides novel insights into the interplay between information, motivation, and behavioral skills to promote safer sexual dual protection practices among female university students. These insights will not only advance our theoretical understanding of the sexual behavior of youths but also inform the development of more comprehensive interventions that address the diverse needs of young people in settings with high HIV burden.

ELIGIBILITY:
Inclusion Criteria:

* Unmarried female students, willing to participate and provide informed consent

Exclusion Criteria:

* Married female students, critically ill and unable to participate in the study.

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1020 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2023-12-20 (Actual)

PRIMARY OUTCOMES:
Dual protection use | at 6 months post-intervention
  Percentage (%) of dual protection use among sexually active participants at last sexual intercourse

SECONDARY OUTCOMES:
Knowledge of safer sexual dual protection behaviors | at 6 months post-intervention
  Percentage (%) of students who have higher knowledge of safer sexual dual protection behaviors
Motivation to practice safer dual protection behaviors | at 6 months post-intervention
  Percentage (%) of students who have a positive attitude toward safer sexual dual protection behaviors
Behavioral skills for practicing safer sexual dual protection behaviors | at 6 months post-intervention
  Percentage (%) of students who have higher self-efficacy for safer sexual dual protection behaviors

CONTACTS AND LOCATIONS:
Overall Officials: Banti N Feyisa, MPH/RH, Principal Investigator — Jimma University, Jimma, Ethiopia; Gurmesa T Debelew, Professor, Study Chair — Jimma University, Jimma, Ethiopia; Zewude B Koricha, Professor, Study Director — Jimma University, Behavioral Science and Society, Jimma, Ethiopia
Locations (1):
- Metu University, Metu, Oromiya, Ethiopia

IPD SHARING:
Plan to Share IPD: Yes
The underlying data supporting the conclusion of this article will be made available to public in an appropriate data repository and under the terms of the CC0 Public Domain Dedication license.
  The specific IPD to be shared will include:
  1. SPSS Datasets: consisting of survey responses of participants' levels of information, motivation, behavioral skills and risky and safer sexual behaviors among female university students at pretest and posttest measures.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The IDP and supporting information will be available immediately following publication and for no end date.
Access Criteria: The IPD and supporting information will be made available to public in an appropriate data repository and under the terms of the CC0 Public Domain Dedication license and can be accessed by everyone who needs it with a responsible use and for further analyses.
URL: https://osf.io/puxgw/

REFERENCES:
- [Background] Teo, T. Structural equation modeling in educational research: Concepts and applications. Chicago: Sense Publishers.2009.
- [Background] SJ, M. A measure of AIDS prevention information, motivation, behavioral skills and behavior. Handbook of sexuality-related measures, 1998, 328-337.
- [Background] HIV/AIDS, J. U. HIV prevention among adolescent girls and young women. Geneva, Switzerland. 2016
- [Background] Fisher JD, Fisher WA, Bryan AD, Misovich SJ. Information-motivation-behavioral skills model-based HIV risk behavior change intervention for inner-city high school youth. Health Psychol. 2002 Mar;21(2):177-86. PMID 11950108
- [Background] Fisher JD, Fisher WA, Williams SS, Malloy TE. Empirical tests of an information-motivation-behavioral skills model of AIDS-preventive behavior with gay men and heterosexual university students. Health Psychol. 1994 May;13(3):238-50. doi: 10.1037//0278-6133.13.3.238. PMID 8055859
- [Background] Fisher JD, Fisher WA, Misovich SJ, Kimble DL, Malloy TE. Changing AIDS risk behavior: effects of an intervention emphasizing AIDS risk reduction information, motivation, and behavioral skills in a college student population. Health Psychol. 1996 Mar;15(2):114-23. doi: 10.1037//0278-6133.15.2.114. PMID 8681919
- [Background] Fisher JD, Fisher WA. Changing AIDS-risk behavior. Psychol Bull. 1992 May;111(3):455-74. doi: 10.1037/0033-2909.111.3.455. PMID 1594721
- [Background] Federal, H. Federal HIV/ AIDS prevention and control office (FHAPCO). HIV/AIDS National Strategic Plan for Ethiopia, 2025. AIDS prevention and control office (FHAPCO), 2021.
- [Background] Demographic, N. Health survey 2011. Central Statistical Agency. Ethiopia ICF International Calverton, Maryland, USA .2012
- [Background] CSA, C. Ethiopia demographic and health survey: key indicators report. Central Statistical Agency, 2016
- [Background] Berer M. Dual protection: more needed than practised or understood. Reprod Health Matters. 2006 Nov;14(28):162-70. doi: 10.1016/S0968-8080(06)28262-4. PMID 17101435
- [Background] Bazargan M, Stein JA, Bazargan-Hejazi S, Hindman DW. Using the information-motivation behavioral model to predict sexual behavior among underserved minority youth. J Sch Health. 2010 Jun;80(6):287-95. doi: 10.1111/j.1746-1561.2010.00503.x. PMID 20573141
- [Background] Bazargan M, Kelly EM, Stein JA, Husaini BA, Bazargan SH. Correlates of HIV risk-taking behaviors among African-American college students: the effect of HIV knowledge, motivation, and behavioral skills. J Natl Med Assoc. 2000 Aug;92(8):391-404. PMID 10992684
- [Background] Aborode AT, Alexiou A, Ahmad S, Yasir Essar M, Chibueze OS, Al-Zahrani Y, Ayomide OE, Batiha GE. HIV/AIDS Epidemic and COVID-19 Pandemic in Africa. Front Genet. 2021 Aug 31;12:670511. doi: 10.3389/fgene.2021.670511. eCollection 2021. No abstract available. PMID 34539728
- See also: Open Science Framework (OSF) repository — https://osf.io/puxgw/
- Available data/document: Individual Participant Data Set: doi.org/10.17605/OSF.IO/SE8M7 — https://osf.io/puxgw/